CLINICAL TRIAL: NCT06616103
Title: Utility of Quantitative Imaging Parameters from Deep Learning-based CT Segmentation in Assessing Hepatic Steatosis and Fibrosis in Chronic Hepatitis B: a Prospective Study Using MRI As the Reference Standard
Brief Title: Quantitative CT Imaging Parameters for Assessing Hepatic Steatosis in CHB
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeongin Yoo, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: CHB prospective MEDIP; RS-2023-00253896 (Other Grant/Funding Number: National Research Foundation of Korea (NRF) grant funded by the Korean government (MSIT))
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Chronic Hepatitis B; Steatosis of Liver; Fibrosis and Cirrhosis of Liver
MeSH Terms: conditions — Hepatitis B, Chronic; Fatty Liver; Fibrosis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: computerized tomography — noncontrast abdominal CT

SUMMARY:
This study aims to evaluate diagnostic performance of CT attenuation parameters acquired using deep learning algorithm in assessing hepatic steatosis and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis B
* no chronic liver disease other than chronic hepatitis B
* Body mass index >= 23

Exclusion Criteria:

* pregnant women
* unable to perform MRI examinations due to claustrophobia or metallic foreign body
* suspicious hepatic malignancy on previous imaging studies
* history of local treatment for hepatic lesions
* history of surgery or catheter insertion of liver or spleen

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B who follow up at Seoul National University Hospital having no history of hepatic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2024-09-26 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance of CT attenuatio parameters in assessing hepatic steatosis and fibrosis | At the time of enrollment
  diagnostic performance of CT attenuatio parameters in assessing hepatic steatosis and fibrosis using MRI-PDFF and MR elastography as reference standards

SECONDARY OUTCOMES:
Consistency between MRI-derived body composition data and CT-derived data | At the time of enrollment
  Consistency between MRI-derived body composition data and CT-derived data using automated 3D organ segmentation algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided